CLINICAL TRIAL: NCT04486469
Title: Efficacy of Physiotherapy Techniques on Irritable Bowel Syndrome
Brief Title: Efficacy of Physiotherapy Techniques on Irritable Bowel Syndrome (IBS). Pilot Study.
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBS Group, Alcalde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBSGroupAlcalde
Record Dates: First submitted 2020-07-19; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 24 patients diagnosed with Irritable Bowel Syndrome
Masking Description: The patients were cited for individual sessions in a close space so they did not know if they all received the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with Irritable bowel syndrome (Experimental): Experimental group is formed with 24 patients diagnosed with IBS treated in the digestive system service of the Virgen de la Arrixaca and Reina Sofía General University Hospitals.
  Interventions: Other: Physical Therapy Group

INTERVENTIONS:
Other: Physical Therapy Group — 1. Performing direct physical treatment on the diaphragm, using stretching, followed by teaching exercises for re-education of the abdomen and diaphragm.
  2. Transcutaneous retrograde electrostimulation: L1-L4 (2hz-10hz) rectangular asymmetric biphasic at the level of the dermatome. From the anterior inferior iliac spine to a pubic symphysis. Second canal from the greater trochanter to the saphenous veins. (30 min). Parameters of this program: 2 Hz and 180ms.
  3. Connective Tissue Massage or Dicke
  4. Massage with direct maneuvers on the abdomen: The direction of the maneuvers will be clockwise. We will perform 6 very slow strokes adding small pressures on the ascending, transverse and descending colon respectively and repeating this maneuver 3 times. (10 minutes)

SUMMARY:
Introduction and State of Question Irritable Bowel Syndrome can be classified as a functional digestive disorder characterized by abdominal pain, bloating, and changes in the frequency and consistency of bowel movements. Recent studies endorse the use of physical therapies for its symptomatic treatment. With the present study investigators wanted to verify the effectiveness of physiotherapy techniques in order to alleviate or eliminate the symptoms of Irritable Bowel Syndrome.

Material and Methods Investigators have carried out an uncontrolled pilot clinical trial in a sample of 24 patients diagnosed with Irritable Bowel Syndrome in two hospitals in the Region of Murcia. Among the measurement tools used, we highlight the use of the IBS-Severity Scale, IBS-QoL, STAI and spirometry tests.

DETAILED DESCRIPTION:
Scope of treatment: From the Digestive System Services, patients who meet the criteria described above, will be referred to the Rehabilitation Services of the Virgin of Arrixaca and Reina Sofía University Hospital, and then, to the physiotherapy unit. At the same time, the researcher will contact these patients to manage the appointments proposed in physiotherapy. The physical treatment to be applied individually has a duration of 40 min per session, establishing a maximum of 8 sessions and a minimum of 3 sessions. This treatment is described below: the first three weeks: (3 days / week)

1. Performing direct physical treatment on the diaphragm, using stretching, followed by teaching exercises for re-education of the abdomen and diaphragm. (20 min):

   A) Direct physical treatment on the diaphragm. It refers to the stretching of the xiphoid and costal portions. With the patient in the supine position and the hips flexed 90º, investigator take advantage of the abdominal-diaphragmatic respiration in its expiratory component to stretch these portions, trying to penetrate with fingertips over the xiphoid and costal edge and maintaining the position with each gain, performing a maximum of 3 winnings.

   B) Abdomino-diaphragmatic reeducation: With the patient in the supine position and the hips flexed 90º, investigator will place the hands in the abdominal area and ask pacient to try to push the hands upwards taking air with the belly. Once the patient have become aware investigator will put up some resistance to the movement. Investigator will avoid possible compensations by controlling the expansion of the rib cage if necessary. Next investigator will ask patient to associate movements of the pelvic scale during breathing. In inspiration, investigator will ask patient to slightly push the sacrum on the stretcher and in ESP, then investigator will ask patient to bring the pelvis back tightening the buttocks as trying to retain defecation. (10min)
2. Transcutaneous retrograde electrostimulation: L1-L4 (2hz-10hz) rectangular asymmetric biphasic at the level of the dermatome. From the anterior inferior iliac spine to a pubic symphysis. Second canal from the greater trochanter to the saphenous veins. (30 min). For this, investigator use the TENS STIM-PRO T-800 device. European Certificate of Conformity (CE 2460). The investigator use program of acupuncture TENS according to the Sjound and Erikson theory of endorphin release, with a neuromodulating objective. Parameters of this program: 2 Hz and 180ms, for 30 min. Investigator should increase the intensity measured in Milli-Amps until it produces contraction for a few seconds, then lower it until the contraction is no longer visible. This therapy can be applied during manual therapy treatment, be it diaphragmatic stretching, abdominal massage and diaphragmatic reeducation.
3. Connective Tissue Massage or Dicke (10 min): Investigator place the patient sitting on the table and ask that the lumbar area and gluteal and sacral area be discovered. Without the help of oils or creams, investigator have to make three strokes with the help of the ulnar edge of the hand and the 3rd and 5th finger. This therapy may arise that the patient has to go to the bathroom before, during or after treatment due to the activation of the renal system through stimulation of the cuti-visceral reflex.
4. Massage with direct maneuvers on the abdomen: It is a massage specially indicated to facilitate intestinal mobility and transit in the large intestine. For its realization investigator can apply creams or oils. The direction of the maneuvers will be clockwise. It is important to apply the not pain rule. Investigator will start with a superficial friction, followed by a spiral massage in the intestinal area. Next, perform 6 very slow strokes adding small pressures on the ascending, transverse and descending colon respectively and repeating this maneuver 3 times. (10min)

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Collaborating patients
* Patients Diagnosed with IBS from the Digestive System Services of the Virgen de la Arrixaca and Reina Sofía Hospital in Murcia in Outpatient Consultations.
* Accept and sign the informed consent
* Degree of Severity in the IBS-Severity index from Moderate to Serious (greater than 175p.)
* Frequency of abdominal pain in 2 out of 10 days in the IBS-SI

Exclusion Criteria:

* Patients with fear or phobia of electricity
* Restrictive diaphragmatic respiratory pathologies in your medical history, either due to neurological or traumatic causes.
* Patients with pacemakers, or diagnosed with heart disease or arrhythmias.
* Presence of developing scars, burns, allergies, wounds or infections in the thigh and lower back application areas.
* undiagnosed pain
* Neoplasms
* Deep venous thrombosis
* Pregnancy

Elimination criteria:

* Worsening of symptoms after abdominal massage
* Failure to attend sessions of 2 or more days followed by treatment

Ages: 36 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
"Change from Baseline IBS-Severity Index at month"- | "up to four weeks"
  The severity questionnaire is divided into 3 sections. The first is the main one, and collects information about the severity. It contains 4 questions, each with a maximum score of 100 using visual analog scales, out of a maximum score of 500.
"Change from Baseline IBS-QoL score at month"- | "up to four weeks"
  It is a self-administered questionnaire, which is usually answered in about 10 min. This consists of 34 items with a value of 5 points each, which collect information on the quality of life of patients affected with IBS. This questionnaire is classified into 8 main areas: dysphoria, interference with activity, body image, health concern, avoidance of food, social relationships, sexual scale and relationships.
"Change from Baseline Trait Anxiety Inventory (STAI) score at month" | "up to four weeks"
  It is divided into two subscales (AE and AR). The AE scale consists of 20 sentences that the subject scores from 0 to 3 and defines how he feels in a "specific moment". Trait anxiety (AR) signals an anxious predisposition to perceive situations as threatening. The AR scale consists of 20 sentences, shows how the subject feels in "general".
"Change from Baseline Simple spirometry parameters at month" | "up to four weeks"
  It is a diagnostic test that allows the detection of respiratory pathologies of an obstructive or restrictive nature, as well as making a differential diagnosis in patients at risk. This device allows investigator to measure the following parameters: Forced Vital Capacity (FVC), Forced Expiration Volume in one second (FEV1), calculate the Tifenneau Index of the examinee by means of the ratio between FEV1 and FVC. It also allows to measure the Peak of Maximum Expiratory Flow (PEF), 25% of FVC flow (FEF25), among others possible.The measurement of these parameters will be carried out with the help of the CONTEC SP10W digital spirometer, with a European Conformity certificate (CE-0123). Electromagnetic Compatibility (EMC): Group I, class B. ¾ Class B (Electromagnetic system, which is marketed for use in a residential environment. Its limits are stricter than industrial devices). Medical devices - covered by directive, 93/42 / EEC. Classification of medical device IIa.

SECONDARY OUTCOMES:
"Change from Baseline Setpoint Abdominal Pain in IBS-Severity Index at month" | "up to four weeks"
  Setpoint of the severity scale that measures the subjective sensation of abdominal pain with a visual scale.
"Change from Baseline Setpoint funcional bloating in IBS-Severity Index at month" | "up to four weeks"
  Setpoint of the severity scale that measures the subjective sensation of bloating
"Change from baseline of bowel movements at month" | "up to four weeks"
  Maximum number of bowel movements in one week

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Gil Alcalde, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Are available for 6 months
Access Criteria: Those researchers who carry out physiotherapy studies for Irritable Bowel Syndrome